CLINICAL TRIAL: NCT07276191
Title: UL Smile - Mobile Application for Oral Health Promotion: Development and Effectiveness Evaluation in Adolescents Living in Portugal: A Randomized Controlled Field Trial
Brief Title: UL Smile: A Mobile Health Application to Promote Oral Health in Portuguese Adolescents
Acronym: UL Smile
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Joana Patrícia, PhD Student Joana Fonseca Costa, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CE-FMDUL202530
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Oral Health Care; Oral Health Behavior Change; Oral Health Self-efficacy
Keywords: Adolescent; Mobile Applications; Oral Health; Health Promotion; MHealth; Health Behavior; Behavior change techniques
MeSH Terms: conditions — Health Behavior | interventions — Telemedicine; Health Education, Dental

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group, cluster-randomized controlled trial. Entire school classes (clusters) are randomly assigned to either the intervention group, which will use the UL Smile mobile application in conjunction with oral hygiene consultation, or the control group, which will receive standard consultation without access to the app. The allocation ratio is 1:1. Cluster randomization at the class level helps prevent cross-contamination between groups. The intervention period lasts approximately three months, with data collected at baseline, 1-month, and 3-month follow-up.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is blinded to group allocation to minimize detection bias. This assessor will perform clinical evaluations (e.g., simplified oral hygiene index, bleeding on probing, DMFT and caries risk assessment) at intermediate and final follow-up points without knowledge of whether participants belong to the intervention or control group. Masking is maintained by using separate investigators for intervention delivery and outcome assessment. Participants, care providers, and the principal investigator are not masked due to the nature of the intervention, which requires active engagement with the mobile app or the standard consultation approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ULSMILE group (Experimental): The intervention arm will receive an oral hygiene consultation supported by the "UL Smile" mobile application, which includes features such as educational videos, brushing guidance, reminders, and motivational messages.Both groups will receive a hygiene kit and be assessed at baseline, 1 month, and 3 months.
  Interventions: Behavioral: Oral Health Behavioral change; Other: MHealth; Other: Oral Health education
- CONTROL group (Active Comparator): The control arm will receive the same oral hygiene consultation without access to the app, using traditional educational materials such as oral cavity models. Both groups will receive a hygiene kit and be assessed at baseline, 1 month, and 3 months.
  Interventions: Behavioral: Oral Health Behavioral change; Other: Oral Health education

INTERVENTIONS:
Behavioral: Oral Health Behavioral change — The app includes goal setting (e.g., brushing twice daily, using floss or interdental brushes), self-monitoring tools (e.g., daily brushing checklists), and individualized feedback provided by oral health professionals through a private section of the app. It also incorporates modeling via instructional videos, direct suggestions for healthy habits, reinforcement through badges and motivational messages upon task completion, and prompts to reinforce key messages and behaviours. These components are based on the Behaviour Change Wheel (BCW) framework and are specifically adapted to adolescent users. Although the control group does not receive a digital behavioural intervention, the oral health education and motivational strategies provided during the hygiene consultation are also informed by the BCW framework, ensuring a consistent theoretical basis across both study arms.
Other: MHealth — Use of a mobile application (UL Smile) to deliver structured oral health content and behavioural strategies directly to adolescents via their smartphones. The app provides personalized and interactive tools, including guided brushing animations, educational videos, and digital reminders. It is designed to be used independently by participants throughout the 3-month study period, integrating oral health promotion into their daily routines in a familiar and accessible format. Participants in the control group do not have access to the mobile application and will receive only the standard oral hygiene consultation.
  Arms: ULSMILE group
Other: Oral Health education — Delivery of evidence-based information on oral hygiene practices, prevention of dental caries and gum disease, use of oral hygiene products, and the impact of diet on oral health. The educational content in the experimental group is delivered through short, age-appropriate videos and visual resources developed in collaboration with oral health and communication experts. Messages are designed to promote awareness, self-efficacy, and long-term habit formation. In the control group, oral health education is provided through a standard hygiene consultation using traditional methods, such as verbal explanations and demonstration with oral cavity models, without the use of the mobile application.

SUMMARY:
This study is part of a doctoral research project in Oral Health Sciences and Technologies, with a specialization in Dental Hygiene, at the Faculty of Dental Medicine, University of Lisbon.

With the advancement of technology, smartphones and mobile applications (apps) have become an integral part of daily life, especially among adolescents and young adults, who are the main users of these devices. In 2023, global app downloads reached an estimated 257 billion, including a growing number of health-related apps, known as Mobile Health or mHealth, and, more specifically, apps targeting oral health.

Oral diseases, such as dental caries and periodontal disease, remain a major public health issue due to their high prevalence and impact on quality of life. Although these conditions are preventable, the adoption and maintenance of healthy behaviors continues to be challenging. Mobile apps may serve as an effective complement to oral health consultations, promoting motivation, adherence to recommendations, and communication with healthcare professionals.

Despite the increasing availability of oral health apps, evidence regarding their effectiveness is still limited. Many of these tools lack scientific rigor and fail to adequately meet users' needs.

In this context, an original Portuguese-language mobile application for promoting oral health was developed, based on current scientific evidence and preliminary exploratory studies involving adolescents and oral health professionals. These studies aimed to identify the most relevant features for this type of tool. The app was designed using the Behaviour Change Wheel (BCW) model, widely recognized for structuring effective behavior change interventions in health.

This mobile app was developed by a multidisciplinary team from the University of Lisbon, involving experts from various faculties, including Psychology, Sciences, Dental Medicine, and Fine Arts. As an original tool, it is not yet available on app stores.

The main aim of this study is to test the effectiveness of this app as a complement to oral health consultations in a population of adolescents living in Portugal, contributing to the advancement of knowledge in this field and to the promotion of more innovative and user-centered clinical practices.

These are the specific objectives of the study:

1. To assess the effectiveness of the app when used as a complement to dental hygiene consultations in relation to several oral health indicators, namely risk of dental caries, gingival inflammation, dental plaque presence, and oral self-care behaviors.
2. To analyze the level of satisfaction and usability of the app's features.

The main hypotheses are:

1. The app will significantly improve oral health indicators, including plaque levels, gingival inflammation, and caries risk, compared to a control group.
2. The app will increase adherence to recommended oral hygiene behaviors (e.g., brushing frequency, interdental cleaning).
3. Adolescents using the app will report higher motivation and self-efficacy for oral self-care.
4. The app will demonstrate high usability and user satisfaction, supporting its potential for broader implementation.

DETAILED DESCRIPTION:
The study is structured into two main phases: the development of the application, followed by a randomized controlled field trial to test its efficacy as a complementary tool to oral hygiene consultations.

The application was developed by a multidisciplinary team including professionals in dentistry, psychology, computer science, and design. It was built based on the Behaviour Change Wheel (BCW) model and integrates evidence-based behavioural change techniques from the Behaviour Change Technique Taxonomy v1 (BCTTv1). The app is designed to be personalized and user-friendly, providing features such as interactive toothbrushing guidance (with audio, video, and 3D animations), educational oral health content, gamified elements (badges and achievements), motivational messages, reminders, and a dedicated section where oral health professionals can upload patient-specific advice. The app adapts to user preferences, such as type of toothbrush (manual or electric), orthodontic appliance use, and daily routines.

The second phase of the study will consist of a parallel-group randomized controlled trial conducted in secondary schools in the Lisbon metropolitan area. The sampling strategy will be multi-stage. First, one or more schools will be selected by convenience, ensuring diversity in student profiles across different academic tracks (e.g., sciences, humanities, arts, and vocational education). Within the selected schools, entire classes will be randomly chosen for inclusion in the study. The principal investigator will visit the classrooms, at the beginning or end of a lesson, coordinated with teachers, to present the study objectives and procedures. Students who meet the inclusion criteria and provide informed assent/consent will be enrolled. For participants aged 18 or older, informed consent will be signed by the individual. For minors, both the adolescent and their legal guardian must sign the assent and consent forms, respectively.

After consent is obtained, participants will complete a baseline questionnaire developed by the investigator. The questionnaire is divided into two sections: the first collects demographic and health information, smartphone operating system details, and app usage frequency; the second assesses oral health knowledge and behaviours. Questionnaire content is based on a literature review and standardised oral health recommendations, and it has been reviewed by a panel of five experts (two dentists, two dental hygienists, and one psychologist).

Class-level randomisation (cluster randomisation) will be used to allocate participants to either the experimental group (which will use the app) or the control group (which will not), in a 1:1 ratio. This approach helps minimise the risk of cross-contamination between groups, as each class is expected to have different schedules and limited interaction with other classes. A total sample of 150 participants (75 per group) will be recruited, allowing for potential attrition, although the calculated minimum sample size was 128 based on an expected effect size of 0.5, a power of 0.80, and a significance level of 0.05.

The study will involve three time points across a 3-month follow-up period. At baseline, participants will undergo a clinical oral health assessment including the Simplified Oral Hygiene Index (OHI-S), Bleeding on Probing Index (BOP), Decayed, Missing and Filled Teeth Index (DMFT), and Caries Risk Assessment using the Cariogram model. All students will then receive an oral hygiene consultation, which includes scaling, polishing, and personalised oral health education. In the experimental group, the app will be used as a support tool during the consultation; in the control group, traditional educational materials (e.g., oral cavity models) will be used. A hygiene kit (manual toothbrush, interdental brush or dental floss and fluoride toothpaste) will be provided to all participants.

Thirty days later, a second clinical assessment (intermediate time point) will be conducted, re-evaluating the OHI-S and BOP. No educational reinforcement will be provided during this visit. A third assessment will take place 60 days after the second, repeating all baseline measurements, including a final questionnaire.

All clinical procedures will take place at the school facilities using portable equipment. The research team will include at least two members: the principal investigator, responsible for group allocation, the oral hygiene consultation, and initial data collection; and a second trained and calibrated examiner who will perform follow-up assessments. The second examiner will be blinded to group allocation to reduce bias. Additional field staff may be present at baseline to support data collection and reduce the time required for clinical observations.

The study will adhere to the principles of Good Clinical Practice and the Declaration of Helsinki. All necessary ethical approvals were obtained, including from the Ethics Committee of the Faculty of Dental Medicine of the University of Lisbon and from the school administrations. Participant anonymity will be strictly preserved: each student will be assigned a unique numerical ID, and only assent/consent forms will contain identifying information. These data will be used solely for contacting participants during follow-up and will be destroyed after data collection is complete.

App usage data will be stored locally on the participants' smartphones and will not be transmitted or shared automatically. Instead, participants will be asked to voluntarily share relevant app data with the research team during the follow-up assessments. This data will be identified only by participant ID numbers.

Data collected throughout the study will be manually entered into SPSS by the principal investigator. Descriptive statistics will be calculated for all variables. Inferential statistics will be applied using appropriate tests with a significance level set at 0.05. To ensure inter-examiner reliability, the Kappa coefficient will be used to assess calibration of the researchers. The Kolmogorov-Smirnov test will be used to assess the normality of the distribution of continuous variables, and the Levene's test will be used to assess homogeneity of variances between groups. Based on the results of these preliminary tests, the decision will be made whether to use parametric or non-parametric tests for further analyses.

If normal distribution is confirmed, comparisons of intraoral indices (e.g., plaque index, bleeding index, caries risk) across the three time points will be performed using the General Linear Model (GLM) Repeated Measures or MANOVA. If normality assumptions are not met, the Friedman test will be applied as a non-parametric alternative. For the analysis of associations between two continuous variables from independent samples, Pearson's correlation coefficient will be used, or Spearman's rank correlation coefficient in the case of non-parametric data.

For bivariate analyses involving independent samples, the t-test for independent means or one-way ANOVA will be applied if assumptions are met. If not, the Mann-Whitney U test or the Kruskal-Wallis test will be used, respectively.

Data management procedures include secure storage of all paper and electronic records. Clinical indices will be recorded using standardised forms and entered into a password-protected database. A 10% random sample will be double-checked against original forms to ensure accuracy. Data validation and cleaning will include range and logic checks. A full data dictionary will be maintained, detailing the origin, coding, and normal range of each variable. Missing data will be assessed for randomness and handled using appropriate imputation techniques or sensitivity analysis.

This project represents a pioneering effort in Portugal to develop and evaluate a theoretically grounded, evidence-based mHealth intervention for adolescent oral health promotion.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 15 and 18 years at baseline.
* Be fluent in Portuguese.
* Have access to a mobile phone or computer/tablet with internet.
* Be willing to participate in the study by providing signed assent/consent. For participants under 18 years old, consent must be signed by a legal guardian.
* Use of the app at least twice during the first month of the study.

Exclusion Criteria:

* Current or previous use of any oral health-related mobile application.
* Not being responsible for their own oral hygiene.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dental caries risk assessed by Cariogram | Baseline and 3-month follow-up
  Evaluation of each participant's individual risk of developing dental caries using the Cariogram tool, a validated computer-based model that considers clinical, behavioural, microbiological, and salivary factors to generate a visual and numerical (percentage) estimation of caries risk. This tool incorporates ten parameters, although it is not mandatory to use all of them, the simplified version can be applied with seven parameters, while still maintaining its clinical usefulness. Each parameter is scored on a scale from 0 to 3, where 0 represents the most favourable condition and 3 the least favourable, contributing differently to the final risk estimation. In the present study, due to resource constraints, Cariogram will be applied without the collection of salivary and microbiological data, acknowledging that this decision may reduce the accuracy of the caries risk assessment.
Gingival inflammation | Baseline, 1-month, and 3-month follow-up
  Measurement of gingival inflammation using the percentage of bleeding sites upon gentle probing, following the Bleeding on Probing Index (BOP), which reflects the presence and severity of gingival inflammation.
Dental Plaque accumulation | Baseline, 1-month, and 3-month follow-up
  The Simplified Oral Hygiene Index (OHI-S) will be used to evaluate soft debris and calculus based on two components: the Debris Index-Simplified (DI-S) and the Calculus Index-Simplified (CI-S). Each component measures the amount of debris or calculus on specific tooth surfaces, allowing the effectiveness of oral hygiene practices to be monitored over time. Teeth will be dried and six specific tooth surfaces examined with a mouth mirror and periodontal probe, each surface scored from 0 to 3 for debris and 0 to 3 for calculus, according to the extent of crown coverage. Component scores will be calculated by averaging the surface scores, and the final OHI-S will be the sum of DI-S and CI-S (range 0-6), categorized as excellent (0), good (0.1-1.2), fair (1.3-3.0), or poor (3.1-6.0) to describe oral hygiene status in the trial.
Oral self-care behaviours | Baseline and 3-month follow-up
  Evaluation of participants' oral hygiene behaviours using a structured self-reported questionnaire administered at two time points (baseline and 3-month follow-up). The questionnaire includes 6 items assessing perceived oral health status, frequency and duration of toothbrushing, use of fluoride toothpaste, use and type of interdental cleaning aids (e.g., dental floss, interdental brushes), and frequency of their use. Questions are closed-ended, using yes/no responses, multiple-choice options, or frequency scales, with a few items allowing open responses for further specification.

SECONDARY OUTCOMES:
Oral health knowledge | Baseline and 3-month follow-up
  Evaluation of participants' knowledge regarding oral health concepts, including causes and prevention of dental caries, correct oral hygiene practices, and the importance of diet and fluoride. Data will by validated self-reported questionnaire administered at two time points. Participants answer to 10 items on a 5-point Likert scale.
App usage frequency (UL Smile) | 3-month follow-up
  Frequency of use of the UL Smile mobile application, as self-reported by participants during the final questionnaire and based on in-app records, including how often brushing animations, videos, or reminders were accessed. Questions are closed-ended, using yes/no responses, multiple-choice options, or frequency scales, with a few items allowing open responses for further specification.
Perceived usefulness of the app | 3-month follow-up
  Participants' perception of the usefulness and impact of the UL Smile app on their oral hygiene behaviours and knowledge is assessed through closed-ended questions, using yes/no responses. Participants are asked whether they found the UL Smile app useful (yes/no). Those who respond affirmatively indicate, via multiple-choice options, which aspects they found beneficial. Options include: motivation to brush teeth at least twice daily, learning correct brushing technique, assistance in maintaining adequate brushing duration, or other specified benefits.
Satisfaction with the mobile application UL Smile | 3-month follow-up
  Overall satisfaction with the UL Smile app, including design, clarity of content, ease of use, and relevance to users' needs, assessed through a satisfaction Likert scale in the final questionnaire, ranging from 0 ("not satisfied at all") to 5 ("very satisfied").

OTHER OUTCOMES:
Suggestions for app improvement | 3-month follow-up
  Open-ended responses collected in the final questionnaire, where participants are invited to provide suggestions to improve the app's content, design, and functionalities, based on their experience during the study. Responses will be thematically analyzed to guide future development.
Qualitative feedback on app usability | 3-month follow-up
  Participants will respond to open-ended questions in the final questionnaire, providing written feedback on their experience using the UL Smile app. They will be asked to identify the feature they liked the most and the one they liked the least, as well as to share any additional comments about what they found helpful or unhelpful. Responses will be thematically analyzed to inform future improvements to the app's content and design.

CONTACTS AND LOCATIONS:
Overall Officials: Sónia Mendes, PhD, Study Director — Faculty of Dental Medicine, University of Lisbon; Luísa Barros, PhD, Study Chair — Center for Research in Psychological Science (CICPSI), University of Lisbon; Carlos Duarte, PhD, Study Chair — Faculty of Sciences, University of Lisbon
Locations (1):
- Faculty of Dental Medicine, University of Lisbon, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa JF, Mendes S. Exploring mobile applications for oral health promotion: a randomized clinical trial. Can J Dent Hyg. Forthcoming. Available from: https://files.cdha.ca/profession/journal/earlyview/CJDH_Early_View--FONSECA--Mobile_apps_for_oral_health.pdf
- [Background] Costa J, Mendes S. Young Portuguese adults' perception of mobile apps for motivation tooral health care. Rev Port Estomatol Med Dent Cir Maxilofac 2024;65(2):59-65. doi:10.24873/j.rpemd.2024.06.1220